CLINICAL TRIAL: NCT07362784
Title: Efficacy And Safety Of Antegrade Uretroscopic Lithotripsy Versus Retrograde Ureteroscopic Lithotripsy In The Treatment Of Upper Ureteric Stones Measuring > 10 mm In Maximum Dimension. A Randomized Comparative Study
Acronym: mm millimeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammad Saad Abdulbaki Hafez Attaby, MD candidate, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAMSU M D 23/2021
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Upper Ureteric Stones
Keywords: flexible ureteroscopy; proximal ureteric stones; laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Antegrade flexible ureteroscopy
  Interventions: Procedure: antegrade flexible ureteroscopy for group A
- group B (Active Comparator): retrograde flexible ureteroscopy
  Interventions: Procedure: retrograde flexible ureteroscopy For group B

INTERVENTIONS:
Procedure: antegrade flexible ureteroscopy for group A — The antegrade approach with this stone size will further prove the superior stone free rate compared with the retrograde approach, widen the indication for the antegrade approach and prove the more favorable perioperative safety profile
  Arms: group A
Procedure: retrograde flexible ureteroscopy For group B — he antegrade approach with this stone size will further prove the superior stone free rate compared with the retrograde approach, widen the indication for the antegrade approach and prove the more favorable perioperative safety profile
  Arms: group B

SUMMARY:
This study aims to assess the efficacy and safety of antegrade flexible ureteroscopic lithotripsy in treating upper ureteric stones >10 mm in maximum dimension and impacted upper ureteric stones irrespective of size in comparison to retrograde ureteroscopic lithotripsy and evaluate feasibility, adverse events, hospital stay and cost benefit of both techniques

DETAILED DESCRIPTION:
Study included 100 patients meeting the inclusion criteria for having an upper urteric stone larger than 10 mm in maximum diameter from the level of pelviureteric junction to upper border of sacroiliac junction and aged ≥18 years. Stones were deemed impacted in case of lack of movement for 1 month on 2 computed tomography scans of urinary tract (CTUT) or non passage of guide wire and / or dye intraoperatively. Exclusion criteria were unresolved urinary tract infection, uncorrected coagulopathy, pregnancy, anatomical abnormalities of the urinary system as horse shoe kidney, pelvic ectopic kidney and ureteric strictures, severe orthopedic malformation hindering prone position or antegrade ureteric access as kyphosis and scoliosis, Pediatric age groups < 18 years, ureteric Stent in place, concurrent renal stones, bladder cancer, upper urothelial tumors or renal tumors. All patients signed an informed consent and were randomized by closed envelop method into 2 groups: group A included 50 patients treated by antegrade flexible URSL and group B included 50 patients treated by retrograde flexible URSL.

Preoperatively, all patients underwent evaluation by medical history, physical examination, laboratory work up including complete blood count (CBC), kidney functions test, liver functions test, hepatitis markers, coagulation profile, completer urine analysis and urine culture with sensitivity. All patients were subjected to imaging studies including pelvi-abdominal ultrasound, plain X-ray of urinary tract and CTUT. Postoperatively, all patient had CBC done a few hours after the procedure, monitored for vital signs and urine color. All patients were assessed for residual stone presence 3 weeks after procedure by CTUT. Stone free status was defined by absence of stone fragment of 4 mm or more in maximum diameter. The primary endpoint was stone free rate. Secondary endpoints were complications, operative time, fluoroscopy time, mean hemoglobin drop, hospital stay and need for auxiliary procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients with upper urteric stone larger than 10 mm in maximum diameter from the level of pelviureteric junction to upper border of sacroiliac junction and aged ≥18 years

Exclusion Criteria:

* unresolved urinary tract infection, uncorrected coagulopathy, pregnancy, anatomical abnormalities of the urinary system as horse shoe kidney, pelvic ectopic kidney and ureteric strictures, severe orthopedic malformation hindering prone position or antegrade ureteric access as kyphosis and scoliosis, Pediatric age groups < 18 years, ureteric Stent in place, concurrent renal stones, bladder cancer, upper urothelial tumors or renal tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
stone free rate | 3 weeks after the intervention
  stone free rate was compared between the 2 arms

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: for 6 months after publication
Access Criteria: access for all requesting urologists via Email of central contact person

REFERENCES:
- [Background] Gokce MI, Akpinar C, Obaid K, Suer E, Gulpinar O, Beduk Y. Comparison of retrograde ureterorenoscopy (URS) and percutaneous anterograde ureteroscopy for removal of impacted upper ureteral stones >10mm in the elderly population. Int Braz J Urol. 2021 Jan-Feb;47(1):64-70. doi: 10.1590/S1677-5538.IBJU.2019.0638. PMID 32840338
- [Background] Elgebaly O, Abdeldayem H, Idris F, Elrifai A, Fahmy A. Antegrade mini-percutaneous flexible ureteroscopy versus retrograde ureteroscopy for treating impacted proximal ureteric stones of 1-2 cm: A prospective randomised study. Arab J Urol. 2020 Aug 23;18(3):176-180. doi: 10.1080/2090598X.2020.1769385. PMID 33029428
- [Background] Mohey A, Abdelfattah AA, Mohammed AE, Marzouk A, El-Dakhakhny AS. Comparative study between antegrade flexible ureteroscopy and reterograde intrarenal surgery in the management of impacted upper ureteric stones 1.5 cm or larger. World J Urol. 2023 Dec;41(12):3731-3736. doi: 10.1007/s00345-023-04672-w. Epub 2023 Nov 3. PMID 37921933

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT07362784/Prot_SAP_ICF_000.pdf